CLINICAL TRIAL: NCT00576784
Title: Multi Center, Open Label Study to Evaluate the Influence of Pioglitazone Treatment Over 6 Months on Metabolic Control in Type II Diabetic Patients Previously Treated With Insulin
Brief Title: Metabolic Effects of Pioglitazone in Type II Diabetic Patients Previously Treated With Insulin
Acronym: PIOswitch
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IKFE Institute for Clinical Research and Development (Other)
Responsible Party: Prof. Thomas Forst, IKFE
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATS-K-013; TAK-PIO-004.2
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Last update posted 2007-12-19 (Estimated); Status verified 2007-12

CONDITIONS: Type 2 Diabetes Mellitus; Insulin Resistance
Keywords: type 2 diabetes; insulin treatment; ß-cell function
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Pioglitazone; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Active Comparator): pioglitazone/glimepiride
  Interventions: Drug: pioglitazone and glimepiride

INTERVENTIONS:
Drug: pioglitazone and glimepiride — switch from any insulin treatment to 30 mg pioglitazone and 3 mg glimepiride.
  Other Names: Actos - pioglitazone; Amaryl - glimepiride

SUMMARY:
The goal of the study is to demonstrate whether a switch from insulin therapy to an oral therapy with pioglitazone/glimepiride will lead to a deterioration of glycemic control (increase in HbA1c by more than 0.5 %) within a 6 month observation period.

DETAILED DESCRIPTION:
To demonstrate that reconverting type 2 diabetic patients from insulin treatment to oral treatment using pioglitazone in combination with or without glimepiride is possible without deterioration of blood glucose control.

Primary aim is to maintain glycaemic control (HbA1c) defined as an increase in HbA1c of not more than 0.5 % after 6 months of treatment (visit 7) compared to baseline HbA1c value (screening visit V1).

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus
* insulin therapy > 1 year
* residual ß-cell function (C-peptide increase in iv glucagon test)
* written informed consent

Exclusion Criteria:

* type 1 diabetes
* oral therapy
* life-threatening disease
* heart failure (NYHA I-IV)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-04; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with an increase in HbA1c by 0.5 % after 6 months of treatment compared to baseline HbA1c value | 6 months

SECONDARY OUTCOMES:
Absolute change of HbA1c Insulin resistance according to minimal model and HOMA-S analysis change of insulin resistance according to minimal model and HOMA-S analysis to baseline first phase insulin response | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- IKFE, Mainz, Germany